CLINICAL TRIAL: NCT07053085
Title: A Randomized Phase II Study of Consolidative Surgery and Radiotherapy With Curative Intent for De Novo Oligometastatic HER2+ Breast Cancer [Ablation and Resection for the Consolidation of Oligometastatic HER2+ Breast Cancer (ARCHER)]
Brief Title: A Study of Surgery and Radiotherapy in People With Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-145
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer; HER2-positive Breast Cancer
Keywords: Consolidative surgery; Radiotherapy; Ablation; Resection; 25-145
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Mastectomy; Radiotherapy; Trastuzumab; pertuzumab; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care arm (Active Comparator): Continuation of first-line systemic therapy will receive the usual approach (drug therapy). Patients will be assigned to the continuation of first-line systemic therapy for an indefinite period per the standard of care. Escalation of systemic-therapy line is at the discretion of the treating physician per standard of care.
  Interventions: Drug: Trastuzumab, Pertuzumab, Paclitaxel, or a combination of these drugs
- Consolidation arm (Experimental): Patients will receive surgery, locoregional radiation therapy, SBRT, and the usual approach
  Interventions: Procedure: Lumpectomy or mastectomy; Radiation: Radiotherapy

INTERVENTIONS:
Procedure: Lumpectomy or mastectomy — Resection of the primary breast tumor (ie. lumpectomy when possible or mastectomy when breast conservation not possible). Surgical resection of the primary breast tumor is to be performed per standard guidelines as applied to localized disease. Breast conserving surgery (ie. lumpectomy) is allowable per patient preference when supported by standard surgical practice. Mastectomy is preferred when breast conservation is declined by the patient, or if breast conservation would otherwise not be feasible in the early-stage setting (e.g. large tumor:breast volume ratio, inability to achieve negative margins with breast conservation, etc)
  Arms: Consolidation arm
Radiation: Radiotherapy — Radiotherapy will be delivered using external beam radiation per the guidelines.Radiotherapy will be delivered using external beam radiation per the guidelines set forth below, targeting two main compartments:
  1. Patients will undergo radiotherapy to the breast/chest wall, and regional nodal basins (including the axilla, supraclavicular fossa and internal mammary chain) per the standard adjuvant approach for locally advanced disease, and
  2. Patient will undergo stereotactic body radiotherapy (SBRT) or similarly-ablative approaches to sites of distant disease, including all observable foci and those that may have since resolved radiographically during systemic therapy
  Arms: Consolidation arm
Drug: Trastuzumab, Pertuzumab, Paclitaxel, or a combination of these drugs — Continue to receive the standard treatment you have already started, which includes trastuzumab, pertuzumab, paclitaxel, or a combination of these drugs. This treatment is not part of the study and will be decided by your regular treating physician.
  Arms: Standard of care arm

SUMMARY:
The researchers are doing this study to see if the combination of surgery, locoregional radiation therapy, SBRT (stereotactic body radiation therapy), and the usual approach is more effective in treating oligometastatic HER2-positive breast cancer than the usual approach alone. The researchers will also study the side effects of the study treatment.

DETAILED DESCRIPTION:
Prior to randomization, patients will receive standard of care first-line systemic therapy as defined by NCCN guidelines (paclitaxel, trastuzumab and pertuzumab at the time of study activation). Following a 3-12 month period without evidence of progression as determined by the treating clinician, patients may be registered and then randomly assigned in 1:1 fashion to one of two study arms. All patients will be followed until progression of disease or 3 years after randomization, whichever comes first. All HER2-directed agents are FDA-approved and administered per standard of care practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Pathologically-confirmed metastatic breast cancer.
* Oligometastatic breast cancer (≤5 discrete metastatic lesions) without CNS involvement; as seen on standard imaging during initial workup and monitoring prior to registration.
* HER2-positive breast cancer per CAP/ASCO guidelines as determined by staff pathologist (any estrogen or progesterone receptor status).
* Based on size and location, all metastatic sites can be safely treated with either SBRT or resection.
* Enrolled at least 3 months (and up to 12 months) after initiation of first-line systemic therapy AND without evidence of progression as determined by treating clinician (whether clinically or radiographically) during this window. (ie. in the judgement of the treating clinician, based on standard evaluations, all known disease must be controlled prior to enrollment).
* ECOG performance status 0-2; KPS 60-100

Exclusion Criteria:

* Any foci of disease progression during initial 3-12 months of first-line systemic therapy (as determined by treating clinician)
* Escalation of systemic therapy line due to progressive disease (i.e. initiated second-line therapy prior to enrollment).
* Comorbidities precluding receipt of radiotherapy, surgery or standard systemic therapy.
* Intracranial or intrathecal/intramedullary spinal disease (ie. CNS involvement is excluded from the study; epidural/vertebral disease is permitted)
* Prior cancer history requiring chemotherapy within the past 10 years (ie. prior cancers are permitted provided no chemotherapy was administered).

Inclusion of Underrepresented Populations

* Individuals of all races and ethnic groups are eligible for this trial. There is no bias towards age or race in the clinical trial outlined. This trial is open to the accrual of men and women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2029-09-17 (Estimated); Study Completion 2029-09-17 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  with PFS defined as the time of randomization to the date of clinical or radiographic disease progression or death (by any cause in the absence of progression).

CONTACTS AND LOCATIONS:
Overall Officials: Lior Braunstein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities ), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org